CLINICAL TRIAL: NCT03515915
Title: Evaluating the Interest of GEP-based Derived Histone Acetylation Score to Identify Myeloma Patients Who Could Benefit From Treatment With HDAC Inhibitor
Brief Title: Use Lay Language. HA Score to Identify Myeloma Patients Who Could Benefit From HDACi Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UF9760
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Patients With Recurrent or Refractory Multiple Myeloma
Keywords: multiple myeloma; HDAC inhibitor; Biomarker
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Panobinostat is a potent oral histone deacetylase inhibitor that alters gene expression through epigenetic mechanisms and inhibits protein degradation. It was recently approved by the US Food and Drug Administration for use in combination with bortezomib and dexamethasone in patients with relapsed multiple myeloma (MM) who have received ≥ 2 prior regimens, including bortezomib and an immunomodulatory drug.

A GEP-based histone acetylation score allowing identification of MM patients with a poor prognosis and who could benefit from HDACi treatment was recently reported(Moreaux et al. BJC. 2013).

Our hypothesis is that the histone acetylation score could be promising to identify MM patients who could benefit from treatment with HDACi and the development of personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory multiple myeloma
* Aged 18 years or more with no upper age limit
* Have signed an informed consent

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Relapsed/refractory multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Response rate 'ORR', PR and better (as per IMWG criteria) of MM patients after treatment with Panobinostat according to histone acetylation score value | 1 day
  Overall Response Response rate 'ORR', PR and better (as per IMWG criteria) of MM patients after treatment with Panobinostat according to histone acetylation score value

SECONDARY OUTCOMES:
Progression free survival will be monitored. | 1 day
  Progression free survival will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: JEROME MOREAUX, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France